CLINICAL TRIAL: NCT05598528
Title: A Multicenter Clinical Study to Explore the Mechanism of Primary Resistance to Third-generation EGFR-TKIs as First-line Treatment in EGFR-positive Advanced NSCLC (PRECISE Study)
Brief Title: Exploring the Mechanism of Primary Resistance to Third-generation EGFR-TKIs as First-line Treatment in EGFR-positive Advanced NSCLC (PRECISE Study)
Acronym: PRECISE
Status: Recruiting | Type: Observational
Sponsor: Second Xiangya Hospital of Central South University (Other)
Collaborators: Xiangya Hospital of Central South University (Other); Shanghai Chest Hospital (Other); West China Hospital (Other); Hunan Cancer Hospital (Other); The Third Xiangya Hospital of Central South University (Other); The First Affiliated Hospital of Xiamen University (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); China-Japan Friendship Hospital (Other); Fudan University (Other); First Affiliated Hospital of Kunming Medical University (Other); Loudi Central Hospital (Other); ZhuZhou Central Hospital (Other); Xiangtan Central Hospital (Other); First People's Hospital of Chenzhou (Other); Yueyang Central Hospital (Other); Yongzhou Central Hospital (Unknown); The First Affiliated Hospital of University of South China (Other); Hunan Provincial People's Hospital (Other); Shaoyang Central Hospital (Unknown); Yiyang Central Hospital (Unknown); Changsha Central Hospital (Other); The first people's hospital of Guiyang (Unknown); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Renmin Hospital of Wuhan University (Other); The First People's Hospital of Changde City (Other); Zhuzhou Second Hospital (Unknown); First Hospital of Changsha (Unknown); Hengyang Central Hospital (Other Government); Huaihua first people's Hospital (Unknown); The First People's Hospital of Xiangtan (Unknown); University of South China Affiliated Nanhua Hospital (Unknown); Xiangxi Autonomous Prefecture People's Hospital (Unknown); People's Hospital of Zhangjiajie (Unknown); Second People's Hospital Of Huaihua (Unknown); Hunan Academy of Traditional Chinese Medicine Affiliated Hospital (Unknown); The Third Hospital of Changsha (Unknown); Xiangya Changde Hospital (Unknown); Changsha County first People's Hospital (Unknown); Hunan Provincial Straight Hospital of Traditional Chinese Medicine (Unknown); Liuyang Hospital of traditional Chinese Medicine (Unknown); Second People's Hospital of Hunan (Other); First Affiliated Hospital of Guangxi Medical University (Other); Guiyang Public Health Treatment Center (Unknown); The Affiliated Bethune Hospital of Shanxi Medical University (Unknown); Hunan University of Traditional Chinese Medicine (Other); Tongji Hospital (Other); The First Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, Fang Wu, Associate Professor, Second Xiangya Hospital of Central South University
Other Study IDs: XYEYY20220928
Record Dates: First submitted 2022-10-25; First posted 2022-10-28 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Lung Cancer, Non-small Cell; EGFR Gene Mutation; EGFR-TKI Resistant Mutation; Primary Resistance; Circulating Tumor DNA
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — 1. The paraffin embeds tumor tissue at diognosis
  2. Peripheral venous blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- EGFR-positive lung patients recieving 3rd generation EGFR-TKIs as first-line therapy: Stage III-IV EGFR-positive lung patients receiving 3rd generation EGFR-TKIs (Osimertinib 80mg/Qd or Almonertinib 110mg/Qd or Furmonertinib 80mg/Qd) as first-line therapy.
  Interventions: Other: Genomic profiles detection; Other: circulating tumor DNA detection

INTERVENTIONS:
Other: Genomic profiles detection — The Paraffin-embedded tumor tissue at diagnosis is collected and assessed by Next- generation gene sequencing
Other: circulating tumor DNA detection — The Plasma at diagnosis and at 1-month treatment are collected and assessed by Next-generation gene sequencing

SUMMARY:
Lung cancer is currently the world's largest malignant tumor for cancer-related deaths with non-small cell lung cancer (NSCLC) accounting for 80%-85%. Epidermal growth factor receptor tyrosine kinase inhibitors (EGFR-TKIs), especially the 3rd-generation EGFR-TKIs have demonstrated strong antitumor effects in EGFR-positive patients.

However, approximately 20% of EGFR-positive were primarily resistant to 3rd generation EGFR-TKIs, i.e., clinical non-response or disease progression in the short term.

This study aimed to clarify the molecular indicators that predict the benefits of 3-rd EGFR-TKIs as first-line therapy in NSCLCpatients with EGFR-positive. Further, to clarify their primary drug resistance mechanisms, which is of great significance for the treatment and clinical decision-making of NSCLC disease.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years;
2. Histological or cytopathological diagnosed NSCLC;
3. According to the American Joint Committee on Cancer (AJCC) eighth edition of the Lung Cancer Staging Manual, the clinical stage is unresectable IIIB-IV or recurrence and metastasis after surgery;
4. At least one measurable lesion can be evaluated according to the Response Evaluation Criteria In Solid Tumours v1.1 (RECIST1.1) criteria;
5. Positive EGFR mutation confirmed by tissue or cytology (pleural fluid, cerebrospinal fluid, etc.);
6. Use of third-generation EGFR-TKIs approved by the NMPA for NSCLC as first-line therapy;
7. Cooperate with the provision of clinicopathological data, imaging data, sample collection, and follow-up required for the research process, and agree to use the test data for subsequent research and product development;
8. Agree to participate in this study and sign an informed consent form.

Exclusion Criteria:

1. Patients who cannot understand the content of the experiment and cannot cooperate, and those who refuse to sign the informed consent form;
2. Pregnant and lactating women;
3. Other malignant neoplastic diseases within 3 years;
4. Patients who have undergone other clinical drug trials;
5. Received systemic anti-tumor therapy within 2 years;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stage IIIB-IV EGFR-positive lung patients receiving 3rd generation EGFR-TKIs (Osimertinib 80mg/Qd or Almonertinib 110mg/Qd or Furmonertinib 80mg/Qd) as first-line therapy.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2021-09-28 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 2 years
  The proportion of patients with a complete response or partial response to treatment according to Response Evaluation Criteria in Solid Tumors (RECIST v1.1)
Progression-free survival (PFS) | 3 years
  Time from the beginning of treatment to the first disease progression (PD) in patients with advanced NSCLC
Differences in genomic profiles of tumor tissues and ctDNA clearance of third-generation EGFR-TKIs sensitive and primary drug-resistant NSCLC. | 3 years
  The patients who don't achieve partial response or progress within 6 months are defined as the primary resistant group. The genomic profiles and ctDNA clearance detected by Next-generation gene sequencing will be compared between the primary drug-resistant group and sensitive-drug group.

SECONDARY OUTCOMES:
Overall survival (OS) | 5 years
  Overall survival (OS) is defined as the duration from the beginning of first-line immunotherapy until death due to any cause. Subjects who are still alive at the end of the study observation period will be censored at the time of last known vital status
Disease Control Rate (DCR) | 3 years
  The proportion of patients with a complete response or partial response or stable desease to treatment according to Response Evaluation Criteria in Solid Tumors (RECIST v1.1)

OTHER OUTCOMES:
The correlation between tumor microenvironment signature and efficacy of 3rd EGFR-TKIs | 3 years
  The baseline paraffin-embedded tissue is collected and assessed by multiplex immunohistochemistry, including T lymphocytes, B lymphocytes, NK lymphocytes, macrophagocyte, and DC cells. And explore the association between tumor microenvironment signature and primary resistance and the efficacy of 3rd EGFR-TKIs during the enrolled observation process.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Oncology, The Second Xiangya Hospital, Central South University, Changsha, Hunan, China